CLINICAL TRIAL: NCT00675740
Title: Effects of Physical Exercise Versus Rosiglitazone on Endothelial Function in Coronary Artery Disease Patients With Prediabetes
Brief Title: Physical Exercise Versus Rosiglitazone in CAD and Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Steffen Desch, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Leipzig 03
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Rosiglitazone; halofantrine; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: rosiglitazone
- 2 (Active Comparator): physical exercise
  Interventions: Behavioral: physical exercise
- 3 (No Intervention): control
  Interventions: Other: control

INTERVENTIONS:
Drug: rosiglitazone — tablets 4 mg daily
  Other Names: Avandia (GlaxoSmithKline)
  Arms: 1
Behavioral: physical exercise — stationary bike 5-6 times a week
  Arms: 2
Other: control — control without intervention
  Arms: 3

SUMMARY:
The aim of this study is to prospectively assess the relative benefits of either treatment with rosiglitazone or physical exercise on endothelial function in patients with impaired fasting glucose or impaired glucose tolerance and coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* impaired fasting glucose or impaired glucose tolerance
* angiographic evidence of coronary artery disease

Exclusion Criteria:

* diabetes mellitus type I or II
* preexisting antidiabetic medication
* unstable angina
* indication for coronary bypass surgery
* significant left main disease
* myocardial infarction within preceding 3 months
* ejection fraction < 40%
* significant heart valve disease
* severe metabolic disorders
* severe disorders in lipoprotein metabolism
* thyroid disorders
* alcohol or drug abuse
* pregnancy
* participation in another trial

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
between-group difference in flow-mediated dilation of the brachial artery | 6 months

SECONDARY OUTCOMES:
relative effects of treatment on parameters of - glucose metabolism - inflammatory plasma markers - markers of endothelial function - cellular markers in muscle and fat biopsies | 6 months